CLINICAL TRIAL: NCT04500886
Title: A Single-center, Open-label, Controlled Clinical Study to Evaluate the Efficacy and Safety of Jinyouli®(PEG-rhG-CSF) for the Recovery of Neutropenia After Chemotherapy in Patients With Hemophagocytic Syndrome
Brief Title: Evaluate the Efficacy and Safety of PEG-rhG-CSF in Patients With Hemophagocytic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-HLH-01
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Hemophagocytic Syndrome
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF group (Experimental): Patients received subcutaneous injection of PEG-rhG-CSF(Jinyouli®)24 hours after the end of chemotherapy, 6mg for patients with body weight ≥ 45kg and 3mg for patients with body weight less than 45kg, once per chemotherapy cycle
  Interventions: Drug: PEG-rhG-CSF
- rhG-CSF group (Active Comparator): Patients received subcutaneous injection of rhG-CSF 24 hours after the end of chemotherapy, 300ug for patients with body weight ≥45kg and 150ug for patients with body weight less than 45kg, Once a day for 3-5 days until the absolute count of neutrophils ≥2×109/L.
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — PEG-rhG-CSF is a sustained-duration form of rhG-CSF, a recombinant methionyl form of human granulocyte colony-stimulating factor (G-CSF), similar to rhG-CSF, PEG-rhG-CSF increases the proliferation and differentiation of neutrophils from committed progenitor cells, induces maturation, and enhances the survival and function of mature neutrophils, resulting in dose-dependent increases in neutrophils.
  Arms: PEG-rhG-CSF group
Drug: rhG-CSF — rhG-CSF can increase the proliferation and differentiation of neutrophils from committed progenitor cells, induces maturation, and enhances the survival and function of mature neutrophils.
  Arms: rhG-CSF group

SUMMARY:
Hemophagocytic syndrome (HPS), also known as hemophagocytic lymphohistiocytosis (HLH), is an immune mediated life-threatening disease. There is no uniform recommendation for salvage treatment of HLH. Based on the results of current clinical trials, the marketing situation of the drug in China, and the use requirements of pegylated recombinant human granulocyte stimulating factor(PEG-rhG-CSF), this study was conducted in patients who received the DEP rescue therapy or dexamethasone combined with VP-16 maintenance therapy. The aim of this study was to evaluate the efficacy and safety of PEG-rhG-CSF(Jinyouli®) for the recovery of neutropenia after chemotherapy in patients with hemophagocytic syndrome.

ELIGIBILITY:
Inclusion criteria：

1. Age ≥ 18 years old, ≤ 70 years old;
2. Patients with hemophagocytic syndrome diagnosed by HLH-2004 diagnostic criteria;
3. Patients who plan to receive rescue treatment or maintenance treatment;
4. The expected survival time is more than 1 month;
5. Patients sign informed consent form.

Exclusion Criteria：

1. Patients who have received bone marrow or hematopoietic stem cell transplantation in the past 3 months;
2. Patients with brain metastases;
3. Patients who are allergic to this product or other biological products derived from genetic engineering E. coli;
4. People with mental or nervous system disorders who cannot cooperate;
5. Pregnant or lactating female patients; women who refuse to accept contraceptive measures ;
6. Researchers determine unsuited to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Duration of grade IV neutropenia | From date of randomization until the date of the study completion，up to 1 year.
  Defined as days when the ANC<0.5×10^9/L occurs to the time when the ANC≥0.5×10^9/L.

SECONDARY OUTCOMES:
The recovery time of neutrophils after chemotherapy | From date of randomization until the date of the study completion，up to 1 year.
  Defined as days when the ANC<2.0×10^9/L occurs to the time when the ANC≥2.0×10^9/L.
Neutrophil dynamic changes | From date of randomization until the date of the study completion，up to 1 year.
  The dynamic changes of neutrophil count were observed after chemotherapy.
Efficacy evaluation of salvage therapy | From date of randomization until the date of the study completion，up to 1 year.
  Complete response (CR) and partial response (PR) rates.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, PHD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, China